CLINICAL TRIAL: NCT02029586
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, 12 Weeks, Therapeutic Exploratory Phase 2 Clinical Study to Evaluate the Safety and Efficacy of MB12066 in Patients With Nonalcoholic Fatty Liver Disease (NAFLD) Except Cirrhosis
Brief Title: Therapeutic Exploratory Phase 2 Study to Evaluate the Safety and Efficacy of MB12066 in Patients With Nonalcoholic Fatty Liver Disease(NAFLD) Except Cirrhosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Yungjin Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB12066_201
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — beta-lapachone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- MB12066 (Experimental)
  Interventions: Drug: MB12066 200mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MB12066 200mg — oral administration, 100mg bid
  Arms: MB12066
Drug: Placebo — oral administration, 100mg bid
  Arms: Placebo

SUMMARY:
This is a controlled study to determine the effectiveness and safety of MB12066 in the treatment of adult patients with Nonalcoholic Fatty Liver Disease(NAFLD) except cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* NAFLD Activity Score(NAS) ≥ 3 (Biopsy-proven)

Exclusion Criteria:

* Alcohol consumption > 20g/day
* Type 1 diabetes or poorly controlled diabetes mellitus (HbA1c ≥ 9%)
* Evidence of other chronic liver disease (e.g. HBsAg positive, anti-HCV positive, autoimmune hepatitis, Wilson's disease, alpha-1 antitrypsin deficiency and etc.)
* ALT, AST > 5X the upper limit of normal
* Serum creatinine ≥ 2mg/dl
* Fibrosis score ≥ 3 according to the NASH CRN fibrosis staging system
* NQO1 T/T type
* Weight loss of more than 5kg within 6 months
* Bariatric surgery within 6 months
* Known alcohol or any other drug abuse in the last five years
* Insulin sensitizers, hepatoprotective agents, anti-oxidants, lipid-lowering agents, drugs induced fatty liver within 1 month

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in hepatic steatosis(%) | baseline, 12 weeks
  The NAFLD Activity Score (NAS) grades NAFLD on liver biopsy based on the individual scoring of steatosis, inflammation and ballooning. The NAS is assessed on a scale of 0 to 8 with higher scores indicating more severe disease and lower scores indicating less severe disease. NAS is obtained by adding steatosis(assessed on a scale of 0 to 3), inflammation (assessed on a scale of 0 to 3) and ballooning (assessed on a scale of 0 to 2).

SECONDARY OUTCOMES:
Proportion of subjects with more than 1 point in total NAFLD Activity Score (NAS) | baseline, 12 weeks
Change in fibrosis score | baseline, 12 weeks
Change in steatosis score | baseline, 12weeks
Change in lobular inflammation score | baseline, 12weeks
Change in ballooning score | baseline, 12weeks
Change in lipid profile | baseline, 4weeks, 8weeks, 12weeks

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Seoul St. Mary's Hospital, Seoul, Banpo-daero Seocho-gu
  - Uijeongbu St. Mary's Hospital, Uijeongbu-si, Cheonbo-ro Gyeonggi-do
  - Seoul National University Hospital, Seoul, Daehak-ro Jongno-gu
  - Keimyung University Donsan Medical Center, Daegu, Dalseong-ro Jung-gu
  - Kyungpook National University Hospital, Daegu, Dongdeok-ro Jung-gu
  - Chung-ang University Hospital, Seoul, Heukseok-dong Dongjak-gu
  - ASAN Medical Center, Seoul, Olympic-ro 43-gil, Songpa-gu
  - Boramae Hospital, Seoul, Sindaebang-dong Dongjak-gu
  - Hanyang University Medical Center, Seoul, Wangsimni-ro Seongdong-gu
  - Severance Hospital, Seoul, Yonsei-ro Seodaemun-gu